CLINICAL TRIAL: NCT05008614
Title: Continuous Erector Spinae Plane Block Versus Thoracic Epidural Analgesia After Thoracotomy: A Randomized Controlled Assessor-blinded Non-inferiority Trial
Brief Title: Comparison of Continuous ESP Versus TEA After Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Susie Yoon, Assistant clinical professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2104-142-1214
Record Dates: First submitted 2021-08-03; First posted 2021-08-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain
Keywords: thoracotomy; lung cancer; interfascial plane block; nerve block
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled assessor-blinded non-inferiority trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor not involved in this study will investigate the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae plane block group (ESP group) (Experimental): Patients receiving continuous unilateral ESP block.
  Interventions:
  Procedure: Ultrasound-guided unilateral ESP block via catheter placement for continuous infusion Drug: Ropivacaine 0.75% Injectable Solution Device: 21-gauge 85 mm perineural catheter, 18-gauge 100 mm stimulator needle (Silverstim, Vygon, Ecouen, France)
  Interventions: Procedure: Erector spinae plane block group
- Thoracic epidural analgesia group (TEA group) (Active Comparator): Patients receiving thoracic epidural analgesia.
  Interventions:
  Procedure: Fluoroscopy-guided thoracic epidural analgesia Drug: Ropivacaine 0.75% Injectable Solution Device: 17-gauge Tuohy needle (FlexTip Plus®, Teleflex Medical, USA)
  Interventions: Procedure: Thoracic epidural analgesia group

INTERVENTIONS:
Procedure: Erector spinae plane block group — Before surgery, an anesthesiologist will perform unilateral ESP block with catheterization under ultrasound guidance in the procedure room.
  Drug: Ropivacaine 0.75% Injectable Solution 0.2% ropivacaine is continuously infused to the erector spinae plane at T5 level via 18G 85 mm perineural catheter (Silverstim, Vygon, Ecouen, France) (basal infusion: 10ml/hr, bolus 5ml, lockout time: 20min)
  Other Names: ESP group
  Arms: Erector spinae plane block group (ESP group)
Procedure: Thoracic epidural analgesia group — Before surgery, an anesthesiologist will perform unilateral ESP block with catheterization under fluoroscopy guidance in the procedure room.
  Drug: Ropivacaine 0.75% Injectable Solution 0.2% ropivacaine is continuously infused to the erector spinae plane at T5 level via 17-gauge catheter (FlexTip Plus®, Teleflex Medical, USA) (Silverstim, Vygon, Ecouen, France) (basal infusion: 3ml/hr, bolus 1ml, lockout time: 20min)
  Other Names: TEA group
  Arms: Thoracic epidural analgesia group (TEA group)

SUMMARY:
This prospective, randomized, assessor-blinded study is designed to evaluate the postoperative analgesic efficacy of the ultrasound-guided continuous erector spinae plane (ESP) block in patients undergoing thoracotomy. We hypothesize that US-guided ESP block is not inferior to thoracic epidural analgesia in terms of postoperative pain control in these patients.

DETAILED DESCRIPTION:
Adult patients undergoing elective unilateral thoracotomy for lung cancer resection are randomly allocated to receive US-guided ESP block (n=31) or thoracic epidural analgesia (n=31). Both procedures are performed prior to surgery. Each patient was assessed by a blinded investigator on postoperative day (POD) 1,2 and 3. The primary outcome is pain severity evaluated by a numeric rating scale (NRS) at POD1.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective thoracotomy for lung cancer
* European Cooperative Oncology Group 0 or 1
* American Society of Anesthesiologists (ASA) physical classification I-III
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* patients with chronic postoperative pain after thoracic surgery
* patients undergoing thoracotomy with chest wall resection
* allergies to anesthetic or analgesic medications
* patients with coagulopathy or who continue to take anticoagulants
* preoperative liver or renal dysfunction
* patients with chronic pain, chronic opioid, analgesic or antidepressant or anticonvulsant use
* Do not understand our study
* Medical or psychological disease that can affect the treatment response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum postoperative pain score at rest on postoperative day 1 | Maximum pain score among the 9 am and 4 pm measurements on postoperative day 1
  pain score measured by the 11-pointed numeric rating scale (0: none/10: worst pain)

SECONDARY OUTCOMES:
Postoperative pain score at rest | 9am/4pm on postoperative day 1, 9am/4pm on postoperative day 2, 9am/4pm on postoperative day 3
  Change in the pain score at rest measured by the 11-pointed numeric rating scale (0: none/10: worst pain) from postoperative day 1 to postoperative day 3
Postoperative pain score at movement | 9am/4pm on postoperative day 1, 9am/4pm on postoperative day 2, 9am/4pm on postoperative day 3
  Change in the pain score at movement measured by the 11-pointed numeric rating scale (0: none/10: worst pain) from postoperative day 1 to postoperative day 3
Change in the total consumption (ml) of patient-controlled analgesia | 9am/4pm on postoperative day 1, 9am/4pm on postoperative day 2, 9am/4pm on postoperative day 3
  total consumption (ml) of epidural or erector spinae plane patient-controlled analgesia
Change in the quality of recovery-15 scale from baseline to postoperative day 3 | Day before surgery and 4pm on postoperative day 3
  measured by the Korean version of the quality of recovery-15
Postoperative pulmonary function test | 3 months after surgery
  measured at outpatient clinic
Incidence of chronic postoperative pain | 3 months after surgery
  measure by the Korean version of the pain DETECT
Incidence of chronic postoperative pain | 6 months after surgery
  measure by the Korean version of the pain DETECT

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea